CLINICAL TRIAL: NCT05344482
Title: A Retrospective Multicenter Study for the Assessment of Effectiveness of Secukinumab as Assessed by Psoriasis Area and Severity Index With Subcutaneous Administration in Adult Patients With Moderate to Severe Plaque Psoriasis in Turkish Population
Brief Title: Evaluation of the Effectiveness of Secukinumab in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457ATR02
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Plaque Psoriasis
Keywords: Secukinumab,; real life,; PASI,; effectiveness,; anti-IL17
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Overall cohort: Secukinumab: Included all the patients treated with secukinumab
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — Included all the patients treated with secukinumab

SUMMARY:
This study was a real-life study which was based on secondary data collection from the electronic or paper medical records from the Dermatology Clinics of the 14 University, Training & Research Hospitals in Turkey. Data were extracted between 02 September 2020 and 29 April 2021.

DETAILED DESCRIPTION:
The study was a retrospective, multicenter, cohort study which was based on data collection at week 4,16 and 52 of secukinumab treatment of moderate to severe plaque psoriasis.

The observational design of the study allowed data collection about secukinumab treatment patterns and clinical and demographic characteristics of plaque psoriasis patients treated with secukinumab for 52 weeks in Turkey. The adults included in the study were treated with secukinumab for 52 weeks. The adults with no available data of PASI scores at specific time points (4, 16 and 52 weeks) and no definite description of treatment cessation were excluded. The study population consisted of adults treated with secukinumab for 52 weeks and adults dropped out before 52 weeks with available data of PASI scores at 4, 16 and 52 weeks and definite description of treatment cessation.

Retrospective data collection from secondary sources (hospital medical records) allowed time and cost saving since description of patients' characteristics, analyses of outcomes of interest and their determinants could be made in a short period of time.

The study consisted of the following periods:

* The index date was the date of initiation of secukinumab
* The study (index) period was between 18 May 2018 to 31 May 2020
* The follow-up (post-index) period was 4,16 and 52 weeks post-index

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of psoriasis
* Age ≥ 18 years at registry baseline.
* Patients with a firm diagnosis of chronic plaque psoriasis for at least 6 months before enrollment
* Secukinumab treatment should be initiated 52 weeks before data collection date
* Moderate to severe plaque psoriasis with PASI score of ≥10 before initiating secukinumab.

Exclusion Criteria:

* Patients diagnosed with others types of psoriasis (pustular psoriasis, erythrodermic psoriasis etc) are excluded.
* Previous exposure to secukinumab or any other biologic drug directly targeting IL-17A or IL-17RA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adults diagnosed as chronic plaque psoriasis with no previous exposure to secukinumab or any other biologic drug directly targeting IL-17A or IL-17RA, whose PASI score was ≥10 before initiation of secukinumab in whom secukinumab had been initiated for at least 52 weeks before data collection date.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients having absolute Psoriasis Area and Severity Index PASI≤3 at week 52 | at week 52
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). Assessment of the effectiveness of secukinumab in subjects with moderate to severe plaque psoriasis was performed based on the percentage of patients who had absolute PASI ≤3 at week 52 in Turkey.

SECONDARY OUTCOMES:
Percentage of patients experiencing a 75% reduction in PASI (PASI75) from baseline | at week 4
  Speed of response to secukinumab according to previous biologic use was demonstrated.
Percentage of patients experiencing a 75% reduction in PASI (PASI90) from baseline | at week 16
  Speed of response to secukinumab according to previous biologic use was demonstrated.
Percentage of PASI 90 responders at week 52 out of PASI 90 responders at week 16 | at week 16 and week 52
  Sustainability rate between week 16 and week 52 which is defined as PASI 90 scores at both milestones was assessed.
Percentage of patients experiencing a 100% reduction in PASI (PASI100) from baseline | at week 52
  PASI 100 responders rate at week 52 was assessed.
Percentage of PASI 90 responders among biologic naive patients vs. biologic experienced patients | at week 52
  Responders rates for biologic naive vs. non-naive patients in terms of PASI 90 at week 52 was evaluated.
Percentage of PASI 90 responder rates at week 52 among smokers vs. non-smokers | at week 52
  Effect of secukinumab treatment response for psoriasis patients (between smokers vs. non-smokers) at week 52 was assessed
Percentage of PASI 75 responder rates among very severe (PASI>20) patients prior the treatment | at week 52
  Effectiveness of secukinumab treatment for very severe ( PASI>20 ) psoriatic patients at week 52 was demonstrated.
Nail psoriasis: percentage of patients experiencing nail psoriasis, number of finger nails involved | at week 52
  Effectiveness of secukinumab in psoriatic manifestations was demonstrated.
Palmoplantar psoriasis: percentage of patients experiencing palmoplantar psoriasis | at week 52
  Effectiveness of secukinumab in psoriatic manifestations was demonstrated.
Scalp psoriasis: percentage of patients experiencing scalp psoriasis | at week 52
  Effectiveness of secukinumab in psoriatic manifestations was demonstrated.
Psoriatic arthritis: percentage of patients experiencing psoriatic arthritis | at week 52
  Effectiveness of secukinumab in psoriatic manifestations was demonstrated.
Percentage of patients who discontinued secukinumab at 52 weeks period | at week 52
  Drug survival as measured by percentage of patients who were persistent secukinumab users, or percentage of patients who discontinued secukinumab at 52 weeks period was reported to describe secukinumab treatment utilization patterns.
Time to discontinuation | at week 52
  Time to discontinuation defined as time from treatment initiation to treatment stop. For patients who stopped secukinumab but re initiated treatment within 90 days after stop date without any other systemic treatment in between will be considered as continued/persistent users.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CAIN457ATR02 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17927